CLINICAL TRIAL: NCT00772174
Title: Double-blind, Randomized, Multicenter, Parallel-Group Study to Evaluate the Effects of Pioglitazone on Metabolic Syndrome in Patients With Type 2 Diabetes Treated With Metformin
Brief Title: Efficacy and Safety Study of Pioglitazone Combined With Metformin on Metabolic Syndrome in Subjects With Type 2 Diabetes
Acronym: PRISMA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Medical Director, Takeda Italia Farmaceutici S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IT-PIO-108; 2006-000725-54 (EudraCT Number); PIOc/LAN07/TIF (Other: Takeda ID); U1111-1115-9278 (Registry Identifier: WHO)
Record Dates: First submitted 2008-10-08; First posted 2008-10-15 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone + Metformin (Experimental)
  Interventions: Drug: Pioglitazone and Metformin
- Metformin (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Pioglitazone and Metformin — Pioglitazone 15 mg, tablets, orally, two-times daily and metformin stable dose, orally, three-times daily for 4 weeks; then increased to pioglitazone 15 mg, tablets, orally, three-times daily and metformin stable dose, orally, three-times daily for up to 20 weeks.
  Other Names: ACTOS®; AD4833
  Arms: Pioglitazone + Metformin
Drug: Metformin — Pioglitazone placebo-matching tablets, orally, two-times daily and metformin stable dose, orally, three-times daily for 4 weeks; then increased to pioglitazone placebo-matching tablets, orally, three-times daily and metformin stable dose, orally, three-times daily for up to 20 weeks.
  Arms: Metformin

SUMMARY:
The purpose of this study was to determine the efficacy of pioglitazone taken with metformin on high-density lipoprotein cholesterol in subjects with Type 2 Diabetes.

DETAILED DESCRIPTION:
Diabetes is none of the most common, chronic diseases worldwide and affects nearly 200 million people. It is the fourth or fifth leading cause of death in developed countries, and it is expected that diabetes will reach epidemic proportions, affecting 333 million people globally by 2025.

The metabolic syndrome is a cluster of the most dangerous cardiovascular risk factors and includes diabetes and pre-diabetes in addition to abdominal obesity, low high-density lipoprotein cholesterol, high triglycerides and hypertension. It is estimated that around a quarter of the world's adult population has metabolic syndrome, and are twice as likely to die and three times as likely to have a heart attack or stroke when compared to people without the syndrome. In addition, non-diabetic people with metabolic syndrome have a fivefold greater risk of developing type 2 diabetes. The clustering of cardiovascular risk factors that typifies the metabolic syndrome is now considered the driving force for a cardiovascular disease epidemic.

Metabolic syndrome has been recently defined by a Consensus Conference of the International Diabetes Federation as a cluster of clinical and laboratory signs characterized by the presence of abnormal deposition of fat tissue in the abdomen and visceral districts, and at least two other clinical and laboratory abnormalities, including altered glucose metabolism or type 2 diabetes and decreased levels of high-density lipoprotein cholesterol. One of the underlying pathophysiological mechanisms of metabolic syndrome is insulin resistance, characterized by an increased glucose output from the liver, and reduced glucose uptake in the muscle and adipose tissue cells. Drugs whose mechanism of action consists of increasing insulin sensitivity in the target tissues are able to reduce the clinical manifestations and consequences of metabolic syndrome.

While each individual component of metabolic syndrome confers an increased risk of cardiovascular-related complications or death, this risk is more pronounced when the syndrome itself is present. The more components of metabolic syndrome are evident, the higher is the cardiovascular mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus.
* Has glycosylated hemoglobin levels between 6.0% and 8.0%.
* Treatment with metformin (2,000 to 3,000 mg daily) for at least 3 months.
* Has reduced high-density lipoprotein cholesterol levels less than 40 mg/dl in males and less than 50 mg/dl in females, irrespective of treatment with statins.
* Has central obesity defined as a waist circumference greater than or equal to 94 cm for men and greater than or equal to 80 cm for females.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.

Exclusion Criteria:

* Has a diagnosis of Type 1 Diabetes Mellitus.
* Required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * other oral antidiabetic drugs than metformin or with insulin in the 3 months preceding study entry.
  * Fibrates
  * Rifampicin
* Has any disease with malabsorption.
* Has acute or chronic pancreatitis.
* Has familial polyposis coli.
* Has a medical history of myocardial infarction, transient ischemic attacks or stroke in the past 6 months.
* Has heart failure as defined by the New York Heart Association classification I-IV.
* Has significant liver impairment, with an alanine aminotransferase level greater than 2.5 the upper limit of normal range.
* Has significant renal impairment, with a serum creatinine level greater than 1.5 mg/dl for men and greater than 1.2 mg/dl for women.
* Has anemia of any etiology (defined as hemoglobin levels less than 10.5 g/dL) or any other hematologic disease.
* Has a diagnosis or suspicion of neoplastic disease.
* History of chronic alcohol or drug abuse.
* Known allergy, sensitivity or intolerance to the study drugs and their formulation ingredients.
* Participation in another trial in the 3 months preceding study entry.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Increase in High-Density Lipoprotein cholesterol levels. | Final Visit.

SECONDARY OUTCOMES:
The change from Baseline in Metabolic Syndrome, as defined by the International Diabetes Federation (aggregate waist circumference, fasting plasma glucose, triglycerides and high-density lipoprotein cholesterol). | Weeks: 8 and 24.
The change from Baseline in Metabolic Syndrome, as defined by the International Diabetes Federation (blood pressure). | At all Visits.
The change from Baseline in Individual Metabolic Parameters (insulin sensitivity and beta-cell function, inflammatory cytokines, adipokines, endothelial functionality). | Weeks: 8 and 24.
Adverse Events. | At all Visits.
The change from Baseline in Laboratory Parameters (hematology, chemistry and urinalysis). | Weeks: 8 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI